CLINICAL TRIAL: NCT03458832
Title: Clinical Trial Readiness to Solve Barriers to Drug Development in FSHD
Acronym: ReSolve
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); FSHD Society (Other); Friends Research Institute, Inc. (Other); Muscular Dystrophy Association (Other); AFM Telethon (Unknown); University of Rochester (Other); Leiden University Medical Center (Other); Dyne Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: STUDY00140842; U01NS101944 (NIH)
Record Dates: First submitted 2018-01-11; First posted 2018-03-08 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2024-08

CONDITIONS: Facioscapulohumeral Muscular Dystrophy
Keywords: muscular dystrophy.; FSHD
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral; Muscular Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Each subject will have approximately 15 mL of blood collected at baseline and month 3 for genetic testing. The month 3 sample will be stored for use as a back-up for any lost samples, or for use in future studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- FSHD-COM: All participants will be asked to undergo FSHD-specific functional rating scale tests and procedures and Electrical Impedance Myography.
  Interventions: Diagnostic Test: FSHD-specific functional rating scale; Device: Electrical Impedance Myography

INTERVENTIONS:
Diagnostic Test: FSHD-specific functional rating scale — The FSHD-COM is composed of disease-relevant functional tasks such as leg function; shoulder and arm function; trunk function, hand function, and balance.
  Other Names: FSHD-COM
Device: Electrical Impedance Myography — EIM is a non-invasive, painless, and fast technique for obtaining information on how a patient's muscle structure is changing. EIM uses a small electrical current to measure the health of the underlying muscle. The patient will be asked to lie down and a trained clinical evaluator will perform testing on 16 total muscles (8 on each side) on your arms and legs.
  Other Names: EIM

SUMMARY:
The primary cause of facioscapulohumeral muscular dystrophy (FSHD), a common adult-onset dystrophy, was recently discovered identifying targets for therapy. As multiple drug companies pursue treatments for FSHD, there is an urgent need to define the clinical trial strategies which will hasten drug development, including creating disease-relevant outcome measures and optimizing inclusion criteria. This proposal will develop two new outcome measures (FSHD-COM and EIM) and optimize eligibility criteria by testing 320 patients across 14 international sites over a period of 24 months.

DETAILED DESCRIPTION:
The overall aim of this study is to hasten drug development for facioscapulohumeral muscular dystrophy (FSHD). Recent breakthroughs in FSHD research have identified the primary disease mechanism as the aberrant expression of a normally silenced gene, DUX4, resulting in a toxic gain-of-function. This disease mechanism is particularly amenable to knock-down of DUX4 using epigenetic strategies or RNA therapies, as well as to other interventions targeting the downstream effects of DUX4 expression. There are many drug companies actively working towards disease-targeted therapies, and two clinical trials either under way now, or planned to start in early Fall 2016. However, meetings with industry, advocacy groups, and FSHD researchers have identified several gaps in the clinical trial arsenal, and clinical trial planning as a major goal for the community. Consequently, there is an urgent need to establish the tools necessary for the conduct of currently planned and expected therapeutic trials in FSHD.

To this end, the researchers propose to develop two novel clinical outcome assessments (COA), a composite functional outcome measure (FSHD-COM) and skeletal muscle biomarker, electrical impedance myography (EIM). In addition, there is broad consensus a better understanding of the relationship of genetic and demographic features to disease progression will be necessary for enumerating eligibility criteria.

The specific aims are to: 1. Determine the multi-site validity of the COAs, 2. Compare the responsiveness of new COAs to other FSHD outcomes and determine the minimal clinically meaningful changes, and 3. establish FSHD cohort characteristics useful for determining clinical trial eligibility criteria. To achieve these aims, the researchers are conducting a multicenter, prospective, 24 months study of 320 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with genetically confirmed FSHD1 or clinical diagnosis of FSHD with characteristic findings on exam and an affected parent or offspring
* Patients with symptomatic limb weakness
* Patients must be able to walk 30 feet without the support of another person or assistance (canes, walking sticks, and braces allowed; no walker).
* If taking over the counter supplements, willing to remain consistent with supplement regimen throughout the course of the study

Exclusion Criteria:

* Patients with cardiac or respiratory dysfunction (deemed clinically unstable, or would interfere with safe testing, in the opinion of the Investigator)
* Patients with orthopedic conditions that preclude safe testing of muscle function
* Patients that regularly use available muscle anabolic/catabolic agents such as corticosteroids, oral testosterone or derivatives, or oral beta agonists
* Patients that have used an experimental drug in an FSHD clinical trial within the past 30 days
* Patients that are pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with FSHD that are seen in the researchers clinic.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2018-03-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
FSHD composite (FSHD-COM) | 24 Months
  The FSHD composite (FSHD-COM) is an 18-item evaluator-administered instrument comprised of individually validated functional motor tasks. The body regions represented match areas of importance identified by patients and include: leg function; shoulder and arm function; trunk function, hand function; and balance. Each item is scored on a 0-4 scale, with 0 representing unaffected/normal performance, and the divisions based on healthy population normative values, or the relative degree of ability to perform the functional task. The total scale has 72 points, with larger weight given to the two most frequently patient-cited areas of functional motor concern - leg function and shoulder and arm function.
Electrical Impedance Myography (EIM) | 24 Months
  EIM is administered using an investigational device manufactured by Skulpt, Inc (Boston, MA) that non-invasively measures the impedance of skeletal muscle over a frequency range between 1 kHz and 10 MHz (Figure 2). The impedance is measured at each frequency by applying low-intensity electrical current (<1 mA) via surface electrodes and measuring the resulting voltage signals using a second set of surface electrodes, converting them into 2 impedance parameters, the resistance and the reactance.

SECONDARY OUTCOMES:
Motor Function Measure (MFM) Domain 1 | 24 Months
  The MFM domain 1 is a validated evaluator administered functional measure for neuromuscular disorders, with 13 items related to standing and transfers.
Facial Function | 24 Months
  The Iowa Oral Performance Instrument (IOPI) is a means to quantify lip, tongue, and buccal strength using a validated tool with published ranges for normative data for lingual measurements.
Reachable Workspace (RWS) | 24 Months
  Subjects are seated in front of a 3D camera and asked to perform a standardized upper extremity movement protocol under the supervision of a study clinical evaluator.
Manual Muscle Testing (MMT) | 24 Months
  Strength testing will be performed using manual muscle testing (MMT) using a hand held force dynamometer.
Force Vital Capacity (FVC) | 24 Months
  The researchers will obtain bedside spirometry including forced vital capacity and forced expiratory volume in 1 second.
Maximum Inspiratory Pressure (MIP) and Maximum Expiratory Pressure (MEP) | 24 Months
  The researchers will obtain maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) using bedside spirometry.
Whole body and regional lean muscle mass (LMM) | 24 Months
  Whole body and regional lean muscle mass (LMM) will be measured via Dual Energy X-Ray Absorptiometry (DEXA).
Severity Scores | 24 Months
  A limited physical exam and strength testing will be used to derive two FSHD clinical severity scores. These severity scores both rank weakness in the face, shoulders, arms, distal, and proximal lower extremities on either a 10 or 15 point scale.
FSHD-Health Inventory (HI) | 24 Months
  The HI is a 15 domain questionnaire designed and based on patient interviews to measure total FSHD health-related quality-of-life, including both motor impairment and the social and emotional impact of FSHD. 116 questions are combined into a total score, the score is transformed onto a percentage scale, with 100 representing maximal disability, and lower scores representing decreasing disability.
Patient-Reported Outcomes Measurement Information System-57 (PROMIS57) | 24 Months
  The PROMIS57 is an instrument developed by the NIH which generates scores for physical function, and the impact of physical limitations on daily life. 57 questions are summed into a total score, which is transformed into a normalized t-score with 50 representing normal, and lower scores representing increasing disability.
The Upper Extremity Functional Index | 24 Months
  This index measures upper extremity dysfunction. 20 questions are combined into a total score, the score is transformed into a normalized score with 80 representing normal, and lower scores representing increasing disability.
The Facial Disability Index (FDI) | 24 Months
  The FDI is a short 5 item questionnaire. The five questions are summed into total score which transformed onto a percentage scale, with 100 representing normal, and lower scores representing increasing disability.
Fall assessment | Total between Month 3 and Month 6 Visit
  Fall assessment will be completed weekly for 3 months after the month 3 visit.
Domain Delta Anchor | 24 Months
  Participants will be asked to complete a self-assessment "domain-delta" questionnaire at 3, 12, 18 and 24-month visits. The purpose of the "domain-delta" questionnaire is to determine each patient's perceived change in their health-related quality-of-life in the last 6-months. This questionnaire will inquire about total health as well as health related to 14 subdomains self-identified as important by patients during development of the FSHD Health Index. Participants indicate their perceived change by answering if an area "is a lot worse", "is a little worse", "there has been no change", "it is a little better", or "it is a lot better" for each subdomain.
Quantitative myometry (QMA) | 24 Months
  Force will be measured on digital myometer, in KG-force.
Muscle Biopsy | 24 Months
  Will be performed on 30 subjects at European and United Kingdom sites only. Participants will undergo one needle muscle biopsy of one lower extremity muscle (Vastus Lateralis (VL), Tibialis Anterior (TA), Medial Gastrocnemius (MG), or Lateral Gastrocnemius (LG)) at any study visit. For each biopsy, approximately three muscle tissue samples will be collected, two samples will be individually flash frozen in liquid nitrogen while the third sample will be put into media for myoblast cell cultures.
Blood biomarkers | 24-Months
  DNA and RNA will be collected at Baseline and 3-month visits. Plasma and serum samples will be collected at every visit (Baseline, 3, 12, 18, and 24-months).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Statland, MD, Principal Investigator — University of Kansas Medical Center; Rabi Tawil, MD, Principal Investigator — University of Rochester
Locations (14):
- United States (8):
  - University of California Los Angeles, Los Angeles, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Rochester Medical Center, Rochester, New York
  - The Ohio State University, Columbus, Ohio
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington
- France (2):
  - Chu De Nice, Nice
  - Institut de Myologie, Paris
- Ludwig-Maximilians-Universität München, München, Germany
- Centro Clinico NeMO, Milan, Italy
- Radboud Unviersity, Nijmegen, Netherlands
- University of College London - Queens Square, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] LoRusso S, Johnson NE, McDermott MP, Eichinger K, Butterfield RJ, Carraro E, Higgs K, Lewis L, Mul K, Sacconi S, Sansone VA, Shieh P, van Engelen B, Wagner K, Wang L, Statland JM, Tawil R; ReSolve Investigators and the FSHD CTRN18. Clinical trial readiness to solve barriers to drug development in FSHD (ReSolve): protocol of a large, international, multi-center prospective study. BMC Neurol. 2019 Sep 10;19(1):224. doi: 10.1186/s12883-019-1452-x. PMID 31506080